CLINICAL TRIAL: NCT05038111
Title: Medical Records Investigation of Whether Perioperative Dexmedetomidine Will Reduce the Duration of Mechanical Ventilation or Hospital Length of Stay in Patients Undergoing Minimally Invasive Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 110006-F
Record Dates: First submitted 2021-08-26; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-03

CONDITIONS: Mechanical Ventilation; Hospital Length of Stay; Minimally Invasive Cardiac Surgery
Keywords: mechanical ventilation; hospital length of stay; dexmedetomidine; Minimally Invasive Cardiac Surgery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Dex: Dexmedetomidine infusion during the perioperative period
  Interventions: Drug: Dexmedetomidine
- Non-Dex: Did not have dexmedetomidine infusion during the perioperative period

INTERVENTIONS:
Drug: Dexmedetomidine — perioperative dexmedetomidine infusion
  Groups: Dex

SUMMARY:
The concept of enhanced recovery after surgery (ERAS) is utilizing in multiple specialties widely. Early tracheal extubation is one of the components of ERAS that enhances postoperative recovery and reduces the length of stay in intensive care unit (ICU).Dexmedetomidine is a highly selective, shorter-acting α2-adrenergic receptor agonist that has both analgesic and sedativeeffects.It was associated with decreased mortality, time to extubation, and hospital length of stay in cardiac surgical patients according to previous studies.The purpose of this study was to investigate the effect of perioperative dexmedetomidine on patients undergoing minimally invasive cardiac surgery(MICS) who were early extubated after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone minimal invasive off-pump coronary artery bypass graft (CABG), valvular surgery or combined procedures at Far Eastern Memorial Hospital, New Taipei City, Taiwan between January 1, 2020 and August 31, 2020.
* Age above 20 y/o

Exclusion Criteria:

* Emergency surgery
* Postoperative mechanical ventilation more than 6 hours
* Extubated in the operating room

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were eligible for inclusion if they had undergone minimal invasive off-pump coronary artery bypass graft (CABG), valvular surgery or combined procedures at Far Eastern Memorial Hospital, New Taipei City, Taiwan between January 1, 2020 and August 31, 2020. Additionally patients were included if they were aged 20 years or older and were excluded if it was emergency surgery, if they had postoperative mechanical ventilation more than 6 hours or if they were extubated in the operating room.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
postoperative mechanical ventilation duration | up to 1 week
  from the time the patient arrived at the ICU until extubation
ICU and hospital length of stay | through admission, up to 1 month

SECONDARY OUTCOMES:
postoperative complications | according to ICD 10 on medical record, daily to discharge, up to 1 month
  atrial fibrillation, bradyarrhythmia, myocardial infarction, cerebrovascular accident, acute renal failure and delirium

CONTACTS AND LOCATIONS:
Overall Officials: Tsung-Hua Yang, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No